CLINICAL TRIAL: NCT01787175
Title: Veterans Affairs Integrated Medication Manager
Brief Title: VA Integrated Medication Manager
Acronym: IMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R18HS017186-03 (AHRQ)
Record Dates: First submitted 2013-01-22; First posted 2013-02-08 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Electronic Health Records
Keywords: Medication Therapy Management; Clinical Decision Support Systems; Medical Informatics; Patient Care Management; United States Department of Veterans Affairs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Medication Manager (Experimental): Experienced providers that participated in the EHR simulations. Half of the providers were assigned to use the new Integrated Medication Manager (intervention) during the simulation. The other half were assigned the VA's CPRS to use (standard EHR). Providers were randomly assigned which system to use.
  Interventions: Other: Integrated Medication Manager
- Standard EHR (No Intervention): Experienced providers that participated in the EHR simulations. Half of the providers were assigned to use the new Integrated Medication Manager (intervention) during the simulation. The other half were assigned the VA's CPRS to use (standard EHR). Providers were randomly assigned which system to use.

INTERVENTIONS:
Other: Integrated Medication Manager — A theory based electronic health record. Half of the provider participants were assigned the IMM to use. The other half were assigned the VA's CPRS EHR to use for the simulation. Providers were randomly assigned to a EHR to use.
  Other Names: IMM
  Arms: Integrated Medication Manager

SUMMARY:
The purpose of this study is to advance the science of healthcare informatics and to improve medication management through the development of a new approach to the electronic medical record called the Integrated Medication Manager (IMM).

DETAILED DESCRIPTION:
In an attempt to address problems patient non-compliance with quality goals barriers to access and integration of health information that impede achievement of treatment goals, the VA is developing a new approach to the electronic medical record. The VA is moving away from the paper-chart metaphor and towards an integrated representation of the patient's status and care process across time. One of the first steps in the development phase has been to explicitly relate patient conditions, therapies, and goals in the domain of pharmacotherapy. This is called Integrated Medication Management and draws on Hollnagel's Contextual Control Model. Providers will be able to plan care and create orders directly in the context of these explicit relationships. This application will be implemented nationwide through a web interface embedded within the existing Computerized Patient Record System (CPRS), the graphical user interface to VA Information Systems (VistA).

Aim 1: Identify cognitive components of providers' therapeutic decision making in the field.

Aim 2. Refine and evaluate the Integrated Medication Manager using simulation studies.

* Aim 2.a. Refine interfaces and logic of the Integrated Medication Manager.
* Aim 2.b. Compare the performance of the Integrated Medication Manager and usual CPRS.

All hypotheses (below) test the use of IMM versus usual electronic medical record (EMR).

* Speed of decision-making will be faster.
* Accuracy of data interpretation (clinical assessment) will be higher.
* Appropriateness of therapeutic plans will be higher.
* Efficiency of gathering information will be higher.
* Common ground measures will be higher.
* Appropriateness of therapeutic plans will be higher when relevant data is outside the usual time horizon.
* Appropriateness of therapeutic plans will be higher when complex associations among patient therapies and goals exist.
* Appropriateness of therapeutic plans will be no lower when relevant data is not captured by the displays of the IMM.
* Appropriateness of therapeutic plans will be higher when highly salient data is not germane to the most important problem.
* Appropriateness of therapeutic plans will be higher when cognitive load is high due to interruptions.

ELIGIBILITY:
Inclusion Criteria:

* Practiced in primary care for at least two years
* Third year residents with two years of residency in internal medicine or family practice
* Do not have to be currently practicing

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Nebeker, MD, MS, Principal Investigator — University of Utah
Locations (1):
- VA SLC Health Care System, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Asch SM, McGlynn EA, Hogan MM, Hayward RA, Shekelle P, Rubenstein L, Keesey J, Adams J, Kerr EA. Comparison of quality of care for patients in the Veterans Health Administration and patients in a national sample. Ann Intern Med. 2004 Dec 21;141(12):938-45. doi: 10.7326/0003-4819-141-12-200412210-00010. PMID 15611491
- [Background] Perlin JB, Pogach LM. Improving the outcomes of metabolic conditions: managing momentum to overcome clinical inertia. Ann Intern Med. 2006 Apr 4;144(7):525-7. doi: 10.7326/0003-4819-144-7-200604040-00012. No abstract available. PMID 16585667
- [Background] Morris AH. Developing and implementing computerized protocols for standardization of clinical decisions. Ann Intern Med. 2000 Mar 7;132(5):373-83. doi: 10.7326/0003-4819-132-5-200003070-00007. PMID 10691588
- [Background] Fox J, Alabassi A, Black E, Hurt C, Rose T. Modelling clinical goals: a corpus of examples and a tentative ontology. Stud Health Technol Inform. 2004;101:31-45. PMID 15537204
- [Background] Xiao Y, Hunter WA, Mackenzie CF, Jefferies NJ, Horst RL. Task complexity in emergency medical care and its implications for team coordination. LOTAS Group. Level One Trauma Anesthesia Simulation. Hum Factors. 1996 Dec;38(4):636-45. doi: 10.1518/001872096778827206. PMID 8976626
- [Background] Phillips LS, Branch WT, Cook CB, Doyle JP, El-Kebbi IM, Gallina DL, Miller CD, Ziemer DC, Barnes CS. Clinical inertia. Ann Intern Med. 2001 Nov 6;135(9):825-34. doi: 10.7326/0003-4819-135-9-200111060-00012. PMID 11694107
- [Background] Nebeker JR, Hurdle JF, Bair BD. Future history: medical informatics in geriatrics. J Gerontol A Biol Sci Med Sci. 2003 Sep;58(9):M820-5. doi: 10.1093/gerona/58.9.m820. PMID 14528038
- [Background] Crosson JC, Stroebel C, Scott JG, Stello B, Crabtree BF. Implementing an electronic medical record in a family medicine practice: communication, decision making, and conflict. Ann Fam Med. 2005 Jul-Aug;3(4):307-11. doi: 10.1370/afm.326. PMID 16046562
- [Background] Hayward RA, Asch SM, Hogan MM, Hofer TP, Kerr EA. Sins of omission: getting too little medical care may be the greatest threat to patient safety. J Gen Intern Med. 2005 Aug;20(8):686-91. doi: 10.1111/j.1525-1497.2005.0152.x. PMID 16050875
- [Background] Tinetti ME, Bogardus ST Jr, Agostini JV. Potential pitfalls of disease-specific guidelines for patients with multiple conditions. N Engl J Med. 2004 Dec 30;351(27):2870-4. doi: 10.1056/NEJMsb042458. No abstract available. PMID 15625341
- [Background] Garg AX, Adhikari NK, McDonald H, Rosas-Arellano MP, Devereaux PJ, Beyene J, Sam J, Haynes RB. Effects of computerized clinical decision support systems on practitioner performance and patient outcomes: a systematic review. JAMA. 2005 Mar 9;293(10):1223-38. doi: 10.1001/jama.293.10.1223. PMID 15755945
- [Background] Shekelle PG. Invited commentary: Implementation of health information technology: an important but challenging field of inquiry. Proc (Bayl Univ Med Cent). 2006 Oct;19(4):313. doi: 10.1080/08998280.2006.11928190. No abstract available. PMID 17106490
- [Background] Weir CR, Nebeker JJ, Hicken BL, Campo R, Drews F, Lebar B. A cognitive task analysis of information management strategies in a computerized provider order entry environment. J Am Med Inform Assoc. 2007 Jan-Feb;14(1):65-75. doi: 10.1197/jamia.M2231. Epub 2006 Oct 26. PMID 17068345
- [Background] Berg CA, Strough JN, Calderone KS, Sansone C, Weir C. The role of problem definitions in understanding age and context effects on strategies for solving everyday problems. Psychol Aging. 1998 Mar;13(1):29-44. doi: 10.1037//0882-7974.13.1.29. PMID 9533188
- [Background] Weir CR. Linking information needs with evaluation: the role of task identification. Proc AMIA Symp. 1998:310-4. PMID 9929232
- [Background] Taatz H. [The problem of the time factor in orthodontic treatment]. Stomatol DDR. 1976 Feb;26(2):102-5. No abstract available. German. PMID 1065968
- [Background] Campbell M, Grimshaw J, Steen N. Sample size calculations for cluster randomised trials. Changing Professional Practice in Europe Group (EU BIOMED II Concerted Action). J Health Serv Res Policy. 2000 Jan;5(1):12-6. doi: 10.1177/135581960000500105. PMID 10787581
- [Background] Miller RH, Sim I. Physicians' use of electronic medical records: barriers and solutions. Health Aff (Millwood). 2004 Mar-Apr;23(2):116-26. doi: 10.1377/hlthaff.23.2.116. PMID 15046136
- [Background] Bradley EH, Bogardus ST Jr, Tinetti ME, Inouye SK. Goal-setting in clinical medicine. Soc Sci Med. 1999 Jul;49(2):267-78. doi: 10.1016/s0277-9536(99)00107-0. PMID 10414834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment 12/2010 to 3/2011 at the Salt Lake City VA and University of Utah health care systems. Simulations took place at either of these locations.
Period: Overall Study
Arm/Group | Integrated Medication Manager | Standard EHR
Started | 30 | 28
Completed | 30 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Half of the providers were assigned to use the new Integrated Medication Manager (intervention) during the simulation. The other half were assigned to use VA's CPRS (standard EHR). Providers were randomly assigned which system to use.
Groups:
- Integration Medication Manager; Standard EHR: Experienced providers that participated in the EHR simulations. Half of the providers were assigned to use the new Integrated Medication Manager (intervention) during the simulation. The other half were assigned the VA's CPRS to use (standard EHR). Providers were randomly assigned which system to use.
- Total: Total of all reporting groups
Arm/Group | Integration Medication Manager | Standard EHR | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 28 | 58
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Amount of Time to Complete Assessment and Plan
Description: Each participant had 10 minutes maximum to review the patient case and write an Assessment and Plan.
Time Frame: 10 minutes
Population: 58 providers were enrolled
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Integrated Medication Manager | Standard EHR
Number analyzed (Participants) | 30 | 28
minutes | 8.5 (1.9) | 8.7 (1.6)
Statistical Analysis 1: Comparison: Integrated Medication Manager; Null hypothesis: Participants will require the same amount of time to complete assessments and plans using either IMM or CPRS. Power calculation: With 2 replications per subject, and assuming an ICC of 0.15, a two-sided alpha 0.05 comparison adjusted for 5 multiple comparisons (adjusted alpha = 0.01), and power of 80%, an N of 32 clinicians was required for each group (32 using IMM, and 32 using CPRS); Test type: Superiority or Other; p = 0.047, Mixed-effects linear model; Difference in time to complete A&P = -17.73, 95% CI 2-sided [-35.24 to -0.23]

2. Primary Outcome: Accuracy of Written Assessment and Plan in Terms of Control and Status
Description: Each participant had 10 minutes maximum to review the patient case and write an Assessment and Plan. The primary outcome evaluated participants' recommendations for treatment of patient conditions. Participants reviewed a total of 10 patient cases and received a score between 0 and 3 points for each issue within each patient case. The final score for each participant was a proportion between 0 and 1. The proportion represented the sum of all points assigned to the participant, divided by the total number of points possible. Higher values on the scale represent greater accuracy of the written assessment and plan.
Time Frame: 10 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Integrated Medication Manager | Standard EHR
Number analyzed (Participants) | 30 | 28
units on a scale | 0.609 [0.581 to 0.637] | 0.569 [0.535 to 0.604]
Statistical Analysis 1: Comparison: Integrated Medication Manager; Null hypothesis: Participants will receive the same scores for assessments and plans completed using either IMM or CPRS. Power calculation: With 2 replications per subject, and assuming an ICC of 0.15, a two-sided alpha 0.05 comparison adjusted for 5 multiple comparisons (adjusted alpha = 0.01), and power of 80%, an N of 32 clinicians was required for each group (32 using IMM, and 32 using CPRS); Test type: Superiority or Other; p = 0.15, Mixed-effects linear model; Value of problem scores for A&P complete = 0.04, 95% CI 2-sided [-0.01 to 0.09]

3. Secondary Outcome: Identification of Planned Monitoring and Follow up Encounters in Assessment and Plan
Description: Each participant had 10 minutes maximum to review the patient case and write an Assessment and Plan. . The secondary outcome evaluated participants' recommendation about future monitoring of patient conditions. Participants reviewed a total of 10 patient cases and received a score of 0 or 1 point for each issue within each case. The final score for each participant was a proportion between 0 and 1. The proportion represented the sum of all points assigned to the participant, divided by the total number of points possible. Higher values on the scale represent a greater proportion of appropriate monitoring recommendations made.
Time Frame: 10 minutes
Measure: Mean (95% Confidence Interval); unit: proportion
Arm/Group | Integrated Medication Manager | Standard EHR
Number analyzed (Participants) | 30 | 28
proportion | 0.505 [0.459 to 0.551] | 0.477 [0.430 to 0.525]
Statistical Analysis 1: Comparison: Integrated Medication Manager; Null hypothesis: Participants will receive the same proportion of acceptable scores for assessments and plans completed using either IMM or CPRS. Power calculation: With 2 replications per subject, and assuming an ICC of 0.15, a two-sided alpha 0.05 comparison adjusted for 5 multiple comparisons (adjusted alpha = 0.01), and power of 80%, an N of 32 clinicians was required for each group (32 using IMM, and 32 using CPRS); Test type: Superiority or Other; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.22 to 2.98]

ADVERSE EVENTS:
Groups:
- Standard EHR: Experienced providers that participated in the EHR simulations. Half of the providers were assigned to use the new Integrated Medication Manager (intervention) during the simulation. The other half were assigned the VA's CPRS to use (standard EHR). Providers were randomly assigned which system to use.
  Integrated Medication Manager: A theory based electronic health record. Half of the provider participants were assigned the IMM to use. The other half were assigned the VA's CPRS EHR to use for the simulation. Providers were randomly assigned to a EHR to use.
Arm/Group | Integrated Medication Manager | Standard EHR
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28

LIMITATIONS AND CAVEATS:
We were not able to evaluate a system-wide deployment of the resulting graphical user interface (GUI) (IMM) in terms of patient outcomes (Aim 3). We were unable to conduct Aim 3, which would have evaluated IMM in a cluster-randomized trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes